CLINICAL TRIAL: NCT06115187
Title: Correlation of Different Ultrasonographic Indices With Clinical Parameters in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Feyza Nur Yucel, Specialist, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: 23-516
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel syndrome; Ultrasound; Echogenicity
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patients with carpal tunnel syndrome
  Interventions: Diagnostic Test: Nerve ultrasound; Diagnostic Test: Nerve conduction studies

INTERVENTIONS:
Diagnostic Test: Nerve ultrasound — Ultrasonographic evaluation of the median nerve at the carpal tunnel and adjacent levels
Diagnostic Test: Nerve conduction studies — Upper extremity nerve conduction studies including median-ulnar sensory and motor responses

SUMMARY:
The aim of this study is to investigate the relationship between different ultrasonographic indices used in patients with carpal tunnel syndrome and clinical parameters.

The main questions it aims to answer are:

* To what extent are the ultrasonographic parameters used in the diagnosis of carpal tunnel syndrome related to the patient's clinical complaints?
* To what extent are the different ultrasonographic parameters used in the diagnosis of carpal tunnel syndrome correlated with each other?

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common entrapment neuropathy and the main mechanism is compression of the median nerve under the transverse ligament at the wrist level. In CTS, neuropathic complaints such as numbness, burning and tingling in the palmar face of the first two fingers, which are the innervation area of the median nerve, and fatigue in the hand are the most common symptoms. In the diagnosis of CTS, the diagnosis is made electrodiagnostically along with typical clinical findings. However, in recent years, ultrasound has become one of the most preferred methods in the diagnosis of CTS because it is non-invasive, rapid and correlates with electrodiagnostic methods. Diameter, cross-sectional area and echogenicity of the median nerve at the carpal tunnel entrance are the most frequently evaluated parameters in ultrasonographic examination. In different studies, it is aimed to increase the power of ultrasonography in the diagnosis of CTS with various indices created in addition to standardized measurements. The most commonly used ultrasonographic indices, which have been shown to be correlated with electrodiagnostic diagnostic methods, are the wrist-forearm median nerve cross-sectional area ratio, the ratio of median nerve cross-sectional area to carpal tunnel area at the carpal tunnel entry level, and echogenicity assessment. Although the relationship of these indexes, which are reported to have sufficient diagnostic sensitivity and specificity, with the patient's clinical complaints is shown on a measurement basis, there is not enough data on the comparison of different formulas and their correlation with the patient's clinical complaints, including neuropathic pain.Based on this, this study aimed to investigate the relationship between ultrasonographic indices used in patients diagnosed with CTS and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with carpal tunnel syndrome based on clinical and electrodiagnostic findings
* Agreeing to participate in the study

Exclusion Criteria:

* Concomitant history of diabetes, systemic inflammatory disease, active infection and malignancy
* Having a disease with neuropathic pain such as polyneuropathy, radiculopathy,multiple sclerosis
* Not agreeing to participate in the study
* History of surgery due to CTS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed CTS
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the carpal tunnel (mm²)
median nerve ultrasound | 3 months
  Median nerve echogenicity at the level of the carpal tunnel (%)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the carpal tunnel inlet (mm²)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the carpal tunnel outlet (mm²)
median nerve ultrasound | 3 months
  Median nerve cross-sectional area measurement at the level of the pronator quadratus (mm²)
median nerve ultrasound | 3 months
  vertical thickness measurement of the median nerve at the level of the carpal tunnel

SECONDARY OUTCOMES:
Visual analog scale | 3 months
  The visual analog scale (VAS) is a validated subjective measure for pain, scored in the 0-10 range (0:no pain; 10: worst pain).
Upper extremity nerve conduction studies | 3 months
  Bilateral median and ulnar sensorimotor latency measurement (msec)
Upper extremity nerve conduction studies | 3 months
  Bilateral median and ulnar motor amplitude measurement (mV)
Upper extremity nerve conduction studies | 3 months
  Bilateral median and ulnar sensory amplitude measurement ( µV)
Upper extremity nerve conduction studies | 3 months
  Bilateral median and ulnar sensorimotor conduction velocity measurement (m/sn)
Self Leeds Assessment of Neuropathic Symptoms and Sign | 3 months
  Self Leeds Assessment of Neuropathic Symptoms and Sign is a 7-question scale used to define pain of neuropathic origin and a score of 12 points or more is in favor of the presence of neuropathic pain.The total score ranges from 0 to 24, and higher scores are associated with an increase in neuropathic complaints.
Boston Carpal Tunnel Questionnaire | 3 months
  he Boston Carpal Tunnel Score is a patient-reported questionnaire that examines symptom severity and overall functional status of patients with carpal tunnel syndrome. Two subscores are calculated: Symptom Severity Scale (SSS) and Functional Status Scale (FSS); SSS score range is 11-55, FSS score range is 8-40 and higher scores indicate worse symptoms or function.
hand grip strength | 3 months
  Grip strength is a measure of muscle strength or the maximum force/tension produced by one's forearm muscles and is measured with a hand dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Assoc.Prof, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Dataset sharing is not planned